CLINICAL TRIAL: NCT01068223
Title: A Single-Center, Single-Dose, Double-Blind, Modified-Double-Dummy, Placebo and Active-Controlled, Randomized, Three-Way, Six-Sequence Cross-Over Study to Investigate the Effect of JNJ-39758979 on Histamine Induced Pruritus in Healthy Male Subjects
Brief Title: A Study To Investigate The Effect of JNJ-39758979 on Histamine Induced Itch in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016609
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Histamine Induced Itch
Keywords: Cetirizine, CR016609

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): A:JNJ-39758979/Placebo #1 Single oral dose of JNJ-39758979 600 mg and Placebo
  Interventions: Drug: A:JNJ-39758979/Placebo #1
- 002 (Placebo Comparator): B: JNJ-39758979 Matching Placebo /Placebo #2 A single dose of 2 different Placebos JNJ-39758979 Matching Placebo and Placebo #2
  Interventions: Drug: B: JNJ-39758979 Matching Placebo /Placebo #2
- 003 (Active Comparator): C:Cetirizine/JNJ-39758979 Matching Placebo Single oral dose of 10mg cetirizine and JNJ-39758979 Matching Placebo
  Interventions: Drug: C:Cetirizine/JNJ-39758979 Matching Placebo

INTERVENTIONS:
Drug: A:JNJ-39758979/Placebo #1 — Single oral dose of JNJ-39758979 600 mg and Placebo
  Arms: 001
Drug: C:Cetirizine/JNJ-39758979 Matching Placebo — JNJ-39758979 Matching Placebo and Placebo #2
  Arms: 003
Drug: B: JNJ-39758979 Matching Placebo /Placebo #2 — A single dose of 2 different Placebos
  Arms: 002

SUMMARY:
The purpose of this study is to investigate the effect of JNJ-39758979 compared to placebo on histamine induced itch in healthy male volunteers.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effect and safety of a single oral dose of JNJ-39758979 on histamine-induced itch and hive in 24 healthy male volunteers. This is a three-treatment, double-blind (neither the volunteer nor the study physician will know the identity of the treatment), cross-over (each volunteer receives all three treatments) study. The study is also randomized, meaning that the order in which treatments are given is determined randomly (by chance, like flipping a coin). The total participation time is approximately 8 to 9 weeks, which includes a screening visit, three treatment periods, two wash-out periods (breaks), and a follow-up visit after the third treatment period. All three treatment periods require a 2-day stay in the clinic. Volunteers will have a histamine test at the screening visit and three times during each treatment period (total of 10 tests). The histamine test consists of an injection of a small amount of histamine solution into the upper layer of the skin, which may cause itchiness, a flare response (redness on the skin) and wheal response (elevated bump in the skin) lasting for 30 to 60 minutes. Volunteers will be blindfolded during the procedure and asked to rate the severity of the itch. The areas of the wheal and flare will be measured by a laser scanner, which will not cause harm to the volunteer. During the treatment periods, volunteers will receive the histamine test on the day before study drug and/or placebo is given and at 2 and 6 hours after study drug and/or placebo is given. During the study, safety evaluations, which will include ECGs (a cardiac function test) and vital signs, will be performed, and side effects will be monitored. Blood and urine samples will be collected at the screening visit, during the first day of each treatment period in the clinic and at the follow-up visit for evaluation. Volunteers will receive single doses of 600mg JNJ-39758979, placebo, and 10mg cetirizine in random order over three treatment periods. The first two treatment periods will be followed by an approximately 14 day wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker or ex-smoker for at least 3 months
* Should generally be in good health
* Must have negative urine alcohol and drug tests
* Must consent to utilize a medically acceptable method of contraception throughout the study and for three months after the last dose of study drug and not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Positive for hepatitis B, hepatitis C, or HIV
* History of drug or alcohol abuse within the past two years
* Known allergies, hypersensitivity, or intolerance to cetirizine (Zyrtec)
* Any confirmed significant reactions against any drug
* Active skin diseases
* History of atopic disease or evidence of allergen sensitization by skin prick testing to common aeroallergens
* Use of antihistamines or antidepressants with antihistamine properties within the last 7 days, prescription medication within the last 14 days or Monoamine oxidase inhibitors (MAOIs) within the last 21 days
* Have received an investigational drug or device within the past 3 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Participant-assessed pruritis score following histamine challenge | at 30 second intervals for the first 5 minutes and then at 1 minute intervals through 10 minutes

SECONDARY OUTCOMES:
To evaluate the effect of single oral dose of JNJ-39758979 (600mg) on histamine-induced wheal and flare in healthy volunteers | at 10 minutes following histamine challenge

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Harrow, United Kingdom